CLINICAL TRIAL: NCT06486662
Title: Safety, Tolerability and Pharmacodynamics of Single and Multiple Ascending Doses of OM-85-IN Versus Placebo in Healthy Volunteers, and Patients With Mild Allergic Asthma Using Nasal Allergen Challenge
Brief Title: A Clinical Study Investigating OM-85-IN Safety and Tolerability in Healthy Volunteers and Mild Allergic Asthma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OM Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BV-2022/11; 2022-503053-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Allergic Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part I -Cohort 1 (Experimental): OM-85-IN low Dose
  Interventions: Drug: OM-85-IN
- Part I -Cohort 1 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part I -Cohort 2 (Experimental): OM-85-IN medium dose
  Interventions: Drug: OM-85-IN
- Part I -Cohort 2 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part I -Cohort 3 (Experimental): OM-85-IN high dose
  Interventions: Drug: OM-85-IN
- Part I -Cohort 3 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part II -Cohort 4 (Experimental): OM-85-IN dose
  Interventions: Drug: OM-85-IN
- Part II -Cohort 4 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OM-85-IN — Participants will receive a Single Ascending Dose (SAD): 1 day single dose treatment and Multiple Ascending Doses (MAD): 16 days multiple dose treatment of OM-85-IN
  Arms: Part I -Cohort 1; Part I -Cohort 2; Part I -Cohort 3; Part II -Cohort 4
Drug: Placebo — Participants will receive a Single Ascending Dose (SAD): 1 day single dose treatment and Multiple Ascending Doses (MAD): 16 days multiple dose treatment of Placebo
  Arms: Part I -Cohort 1 Placebo; Part I -Cohort 2 Placebo; Part I -Cohort 3 Placebo; Part II -Cohort 4 Placebo

SUMMARY:
This study will assess the safety and tolerability of OM-85-IN compared to placebo in healthy volunteers and mild asthmatic patients

DETAILED DESCRIPTION:
This study is a double-blind, randomised, placebo-controlled, single and multiple ascending doses, parallel group design study that aims to assess the safety and tolerability of OM-85-IN compared to placebo in healthy volunteers and mild asthmatic patients

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 55 years. Women will be considered for inclusion if they are:

   * Not pregnant, as confirmed by pregnancy test, and not breastfeeding.
   * Of non-childbearing potential, or
   * Of childbearing potential and using a highly effective method of contraception .
2. Body mass index (BMI) ≥18 and ≤32 kg/m2.
3. Part II : History of mild asthma that is well controlled with Step 1 treatment according to GINA guidelines 2023 for at least 12 months prior to the Screening Visit, i.e., a history of respiratory symptoms such as wheeze, shortness of breath, chest tightness, cough, and limitation of airflow induced by aeroallergens.
4. Part II: Forced Expiratory Volume in the first second (FEV1) ≥80% of predicted at Screening Visit.
5. Part II : Positive skin prick test to common aeroallergens such as tree, weed, grass or house dust mites within 12 months prior to the Screening Visit
6. Part II : Production of adequate sputum with ≥2 x 105 total non-squamous cells within 12 months to 2 weeks prior to V1A (Day -8)
7. Part II : Positive reaction to Nasal Allergen Challenge (NAC) within 12 months to 2 weeks prior to baseline

Exclusion criteria:

1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, lung function or electrocardiogram (ECG) at Screening Visit, which, in the opinion of the Investigator, may either put the subject at risk because ofvparticipation in the study or may influence the results of the study, or the subject's ability to participate in the study."
2. Use of prohibited medication prior to study enrolment
3. Part II - Long-term, daily treatment with inhaled corticosteroids.
4. Part II - Exacerbation of asthma defined according to the GINA guideline 2023 as a progressive increase in symptoms of shortness of breath, cough, wheezing or chest tightness and progressive decrease in lung function, i.e., they represent a change from the patient's usual status that is sufficient to require treatment changes within 1 month prior to the Screening Visit.
5. Part II - Concomitant allergies to seasonal aeroallergens which are anticipated to be or become active during study participation.
6. Known allergy to IMP active substance and/or excipients or the challenge agent components.
7. Specific immunotherapy in the past 3 years before Baseline, ongoing treatment with any specific immunotherapy or plan to receive such treatment during study participation.
8. Previous or ongoing treatment with other bacterial lysates and/or probiotics (dietary supplements, medicinal products and/or other health products) within 30 days before Baseline.
9. Patients with pathological skin modifications in the test area (e.g., acute or chronic eczema or skin infections), with disturbed skin reactivity (e.g., hyperkeratosis, ichthyosis, urticaria factitial), or with acute, generalized hypersensitivity reactions.
10. Participation in any other clinical study within 30 days prior to Screening.
11. Past or present disease, which as judged by the Investigator, may affect the outcome of this study.
12. Positive serology test for hepatitis B surface antigen (HBsAg), hepatitis B core antibodies, hepatitis C virus antibodies (HCV-Ab) or human immunodeficiency virus (HIV) antibody at Screening Visit
13. History or presence of clinically significant hypertension
14. History of anaphylactic shock, generalised exanthema, angioedema or hypotension caused by the allergen used for NAC, or any medicinal product in the past.
15. History of drug or alcohol abuse in the past 12 months.
16. Current smokers or ex-smokers for less than 6 months or more than 10 pack years. Current vapers (users of e-cigarette products) or ex-vapers for less than 6 months.
17. Part II : Negative reaction in the baseline NAC

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events (TEAEs) (including clinically relevant findings from nasal inspection) | 28 days

SECONDARY OUTCOMES:
Part II : Mean difference of Total Nasal Symptom Score (TNSS points) before and after treatment defined as the arithmetic mean of TNSS collected from pre-Nasal Allergen Challenge (NAC) to 6 hours post-NAC | 28 days
Part II : Area under the curve (AUC)0-6 hours of Total Nasal Symptom Score (TNSS points) after NAC before and after treatment | 28 days
Part II : Mean difference of nasal flow by rhinomanometry (Pascal) before and after treatment defined as the arithmetic mean of TNSS collected from pre-Nasal Allergen Challenge (NAC) to 6 hours post-NAC | 28 days
Part II : Area under the curve (AUC)0-6 of nasal flow by rhinomanometry (Pascal) after NAC before and after treatment | 28 days
Part II : Mean difference in fractional exhaled nitric oxide (FeNO) before and after treatment and NAC | 28 days
Part II : Mean difference on mannitol dose resulting in ≥15% fall in FEV1 from baseline or ≥10% incremental fall in FEV1 between consecutive mannitol doses after NAC before and after treatment | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Fraunhofer Institute For Toxicology And Experimental Medicine ITEM, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No